CLINICAL TRIAL: NCT06745076
Title: A Multicenter Study PRECISE-HL: Personalized Reduction of Chemotherapy Intensity Through ctDNA Evaluation in Advanced Hodgkin Lymphoma
Brief Title: Personalized Reduction of Chemotherapy Intensity Through ctDNA Evaluation for the Treatment of Patients With Advanced Hodgkin Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RG1124935; NCI-2024-09815 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20689 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2024-12-13; First posted 2024-12-20 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-12

CONDITIONS: Advanced Hodgkin Lymphoma; Classic Hodgkin Lymphoma; Lugano Classification Stage III Hodgkin Lymphoma AJCC v8; Lugano Classification Stage IV Hodgkin Lymphoma AJCC v8
MeSH Terms: interventions — Specimen Handling; Dacarbazine; Doxorubicin; Nivolumab; Magnetic Resonance Spectroscopy; Vinblastine; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Arm I (MRD negative) (Experimental): CYCLES 1-2: Patients receive nivolumab IV, doxorubicin IV, vinblastine IV and dacarbazine IV on days 1 and 15 of each cycle. Cycles repeat every 28 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity. Patients then undergo MRD testing.
  CYCLES 3-4: Patients receive nivolumab IV, doxorubicin IV, vinblastine IV and dacarbazine IV on days 1 and 15 of each cycle. Cycles repeat every 28 days for up to 2 cycles in the absence of disease progression of unacceptable toxicity.
  CYCLES 5-6: Patients receive nivolumab IV on days 1 and 15 of each cycle. Cycles repeat every 28 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity.
  Patients undergo echocardiography or MUGA scan, PET/CT scan, questionnaire and blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Dacarbazine; Drug: Doxorubicin; Procedure: Echocardiography Test; Procedure: Multigated Acquisition Scan; Biological: Nivolumab; Procedure: Positron Emission Tomography; Drug: Vinblastine; Other: Questionnaire
- Arm II (MRD positive) (Experimental): CYCLES 1-2: Patients receive nivolumab IV, doxorubicin IV, vinblastine IV and dacarbazine IV on days 1 and 15 of each cycle. Cycles repeat every 28 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity. Patients then undergo MRD testing.
  CYCLES 3-6: Patients receive nivolumab IV, doxorubicin IV, vinblastine IV and dacarbazine IV on days 1 and 15 of each cycle. Cycles repeat every 28 days for up to 4 additional cycles (total of 6 cycles) in the absence of disease progression or unacceptable toxicity.
  Patients undergo echocardiography or MUGA scan, PET/CT scan, questionnaire and blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Dacarbazine; Drug: Doxorubicin; Procedure: Echocardiography Test; Procedure: Multigated Acquisition Scan; Biological: Nivolumab; Procedure: Positron Emission Tomography; Drug: Vinblastine; Other: Questionnaire

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Drug: Dacarbazine — Given IV
  Other Names: 4-(Dimethyltriazeno)imidazole-5-carboxamide; 5-(Dimethyltriazeno)imidazole-4-carboxamide; Asercit; Biocarbazine; Dacarbazina; Dacarbazina Almirall; Dacarbazine - DTIC; Dacatic; Dakarbazin; Deticene; Detimedac; DIC; Dimethyl (triazeno) imidazolecarboxamide; Dimethyl Triazeno Imidazol Carboxamide; Dimethyl Triazeno Imidazole Carboxamide; dimethyl-triazeno-imidazole carboxamide; Dimethyl-triazeno-imidazole-carboximide; DTIC; DTIC-Dome; Fauldetic; Imidazole Carboxamide; Imidazole Carboxamide Dimethyltriazeno; WR-139007
Drug: Doxorubicin — Given IV
  Other Names: Adriablastin; Hydroxydaunomycin; Hydroxyl Daunorubicin; Hydroxyldaunorubicin
Procedure: Echocardiography Test — Undergo echocardiography
  Other Names: EC; Echocardiography
Procedure: Multigated Acquisition Scan — Undergo MUGA scan
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Biological: Nivolumab — Given IV
  Other Names: ABP 206; BCD-263; BMS 936558; BMS-936558; BMS936558; CMAB819; MDX 1106; MDX-1106; MDX1106; NIVO; Nivolumab Biosimilar ABP 206; Nivolumab Biosimilar BCD-263; Nivolumab Biosimilar CMAB819; ONO 4538; ONO-4538; ONO4538; Opdivo
Procedure: Positron Emission Tomography — Undergo PET scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Drug: Vinblastine — Given IV
  Other Names: Vincaleucoblastine; VLB
Other: Questionnaire — Complete questionnaire

SUMMARY:
This phase II trial tests how well personalized reduction of chemotherapy (nivolumab, doxorubicin, vinblastine and dacarbazine) based on circulating tumor deoxyribonucleic acid (ctDNA) evaluation works for treating patients with Hodgkin lymphoma that may have spread from where it first started to nearby tissue, lymph nodes, or distant parts of the body (advanced). Chemotherapy drugs, such as nivolumab, doxorubicin, vinblastine and dacarbazine, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Many types of tumors tend to lose cells or release different types of cellular products including their DNA, which is referred to as ctDNA, into the bloodstream before changes can be seen on scans. Health care providers can measure the level of ctDNA in blood or other bodily fluids and, based on the result, assign patients to a reduced number of chemotherapy treatments or the standard number of chemotherapy treatments. Using ctDNA to assign a personalized reduction of chemotherapy may be effective in treating patients with advanced Hodgkin lymphoma.

DETAILED DESCRIPTION:
OUTLINE:

CYCLES 1-2: Patients receive nivolumab intravenously (IV), doxorubicin IV, vinblastine IV and dacarbazine IV on days 1 and 15 of each cycle. Cycles repeat every 28 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity. Patients then undergo measurable residual disease (MRD) testing.

Patients who are MRD negative are assigned to Arm I and patients who are MRD positive are assigned to Arm II.

ARM I:

CYCLES 3-4: Patients receive nivolumab IV, doxorubicin IV, vinblastine IV and dacarbazine IV on days 1 and 15 of each cycle. Cycles repeat every 28 days for up to 2 cycles in the absence of disease progression of unacceptable toxicity.

CYCLES 5-6: Patients receive nivolumab IV on days 1 and 15 of each cycle. Cycles repeat every 28 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity.

ARM II:

CYCLES 3-6: Patients receive nivolumab IV, doxorubicin IV, vinblastine IV and dacarbazine IV on days 1 and 15 of each cycle. Cycles repeat every 28 days for up to 4 additional cycles (total of 6 cycles) in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 1 year then periodically for up to 5 years.

Patients undergo echocardiography or MUGA scan, position emission tomography (PET)-computed tomography (CT) scan, questionnaire and blood sample collection throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Classical Hodgkin lymphoma without prior systemic therapy, stage 3 or 4. Corticosteroids for symptom relief are allowed
* Measurable disease per Lugano criteria
* Patients must be appropriate candidates for 6 cycles of combination chemotherapy including an anthracycline
* No evidence of active central nervous system lymphoma
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Absolute neutrophil count (ANC) ≥ 500/mm^3. Growth factor and/or transfusion support is permissible to stabilize participant prior to study treatment if needed. There is no lower limit to cytopenias if related to bone marrow involvement or underlying Hodgkin lymphoma
* Platelets ≥ 50,000/mm^3 (without transfusion or growth factor support). Growth factor and/or transfusion support is permissible to stabilize participant prior to study treatment if needed. There is no lower limit to cytopenias if related to bone marrow involvement or underlying Hodgkin lymphoma
* Hemoglobin ≥ 8 g/dL. Growth factor and/or transfusion support is permissible to stabilize participant prior to study treatment if needed. There is no lower limit to cytopenias if related to bone marrow involvement or underlying Hodgkin lymphoma
* Serum creatinine < 1.5 x upper limits of normal (ULN) or creatinine clearance greater than 30/ml per minute by Cockcroft Gault formula
* Total bilirubin ≤ 1.5 times upper limit of normal OR direct bilirubin ≤ ULN for participants with total bilirubin levels > 1.5 × ULN). Patients with Gilbert Syndrome and direct bilirubin < 1.5 x ULN or confirmatory UGT1A1 testing are allowed to enroll
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 times upper limit of normal (≤ 5 × ULN for participants with liver involvement)
* Patients must be age 18 or older
* All patients must be informed of the investigational nature of this study and have given written consent in accordance with institutional and federal guidelines
* Patients must be anticipated to complete all planned study therapy
* Male patients must agree to use an adequate method of barrier contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy
* Female patients of childbearing potential must have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Female patients of childbearing potential must be willing to use 2 methods of birth control or be surgically sterile or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year

Exclusion Criteria:

* Patients known positive for HIV or infectious hepatitis type B or C with a detectable viral load may not participate. Hepatitis B/C, and HIV testing are not required at screening unless mandated by local health authority.

  * Patients living with HIV, on anti-viral treatment and undetectable viral load are allowed
  * Patients with positive hepatitis (hep) B core antibody are allowed on study with an undetectable viral load and appropriate prophylaxis
  * Patients with positive hepatitis C antibody are allowed with undetectable viral load
* Pregnant or nursing women. Men or women of reproductive potential may not participate unless they have agreed to use an effective contraceptive method
* Patients with other prior malignancies except for adequately treated basal cell carcinoma, squamous cell carcinoma of the skin, breast or cervical cancer in situ, or other cancer from which the patient has been disease-free for 2 years or greater, unless approved by the principal investigator
* Patients who have other medical conditions that would contraindicate treatment with aggressive chemotherapy (including active infection, uncontrolled hypertension, congestive heart failure, unstable angina pectoris, or myocardial infarction within the past 6 months, uncontrolled arrhythmia, severe pulmonary disease or requirement of supplemental oxygen)
* Active ischemic heart disease (eg. myocardial infarction within 6 months) or congestive heart failure (eg. left ventricular ejection fraction < 50%)
* Concurrent use of other anti-cancer agents or experimental treatments
* Known current or prior autoimmune disease with the exception of vitiligo. Patients with a history of autoimmune thyroid disease on a stable dose of thyroid hormone are also allowed
* Active or prior history of pneumonitis/interstitial lung disease that required corticosteroids
* Current use of supplemental oxygen
* Is known to have received a live vaccine or live-attenuated vaccine within 30 days prior to the first dose of trial treatment. Other non-live or live-attenuated vaccines (eg. COVID, Influenza) are allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2025-03-06 (Actual); Primary Completion 2032-01-03 (Estimated); Study Completion 2033-01-03 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) in patients with undetectable minimal residual disease (MRD) after 2 cycles of treatment | At 1 year

SECONDARY OUTCOMES:
PFS in MRD positive patients after 2 cycles of treatment | At 1 year
PFS in the overall cohort | At 2 years
Best response | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Lynch, MD, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (3):
- United States (3):
  - Washington University in St. Louis, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No